CLINICAL TRIAL: NCT01566812
Title: BReast Feeding Attitude and Volume Optimization (BRAVO) Trial: A Randomized Breast Feeding Optimization Experiment
Brief Title: Effect of Breastfeeding Optimization on Early Vascular Development
Acronym: BRAVO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Collaborators: CEEBM (Unknown); Julius Center (Other); Budi Kemuliaan Hospital (Unknown)
Responsible Party: Principal Investigator, Nikmah Salamia Idris, Dr., Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BRAVO_trial
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Breast Feeding; Cardiovascular Diseases
Keywords: Breast Feeding; Cardiovascular Risk
MeSH Terms: conditions — Breast Feeding; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Breast feeding optimization (Experimental)
  Interventions: Behavioral: Breast feeding optimization; Behavioral: Usual care
- Usual/routine care (Active Comparator)
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Breast feeding optimization — Breast feeding optimization program extends from late pregnancy period to 6 months after birth. Prenatal intervention consists of individual and group counseling/education; perinatal intervention consists of in-hospital lactation support; postnatal intervention consists of home visit, counseling session, reminding telephone call and bulk SMS, special counseling for working mothers, breast pump rental, occupational-related support
  Arms: Breast feeding optimization
Behavioral: Usual care — Usual care applied in the hospital

SUMMARY:
This study aims to find out whether breast feeding optimization will increase breast feeding rates and to evaluate its effect on cardiovascular risk and general health of children.

DETAILED DESCRIPTION:
Breast feeding is suggested to give many benefits for babies and there are some initial prove that it might affect their future health, including the development of cardiovascular diseases. In Indonesia, breast feeding rates are very low, while there is a strong upsurge of cardiovascular disease. In this study, we propose to randomly allocate pregnant Indonesian women who plan to give breast feeding for no more than two months, to either care as usual or to a breast feeding empowerment program lasting to 6 months post partum. At the age of one year, all randomized offspring will undergo non-invasive echographic aortic vascular measurements and cardiovascular risk profiling. Measurements for assessing children's general health status will also be performed, including growth monitoring, repeated lung function test, and microbiomic sampling.

ELIGIBILITY:
Inclusion criteria

* Plan to breast feed for ≤2 months
* Residing in vicinity ≤ 5 km from the hospital/agree to comply to health visit schedule
* Telephone communication is possible
* No known HIV or active tuberculosis in mother
* Uncomplicated pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2012-06; Primary Completion 2018-02 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular risk | 5 years
  Abdominal aortic/carotid intima media thickness, distensibility, elastic modulus; pulse wave velocity, stiffness index, blood pressure; echocardiography: ejection fraction (%), fractional shortening (%), TAPSE (cm), cardiac index (L/min/m2), LV mass (grams)
Breastfeeding habits | 1 years
  Breastfeeding practice: Y/N, night/day, frequency (time interval between breastfeeding, e.g 2 hours) Supplementary formula: frequency/day, volume per feeding Complementary feeding: Y/N, type of foods; frequency/day Employer and employee satisfaction

SECONDARY OUTCOMES:
Child growth | 5 years
  Body weight, height, head circumference, abdominal circumference
Lung function | 5 years
  Resistance, compliance, time constant, FVC (liters), FEV1 (liters) measured by spirometry
Microbiome | 1 years
  Infant nasopharyngeal & oral flora, digestive tract/feces flora, maternal oropharyngeal evaluated using PCR and culture.
Development | 5 years
  Bayley Infant Scales, IQ
Illness | 1 year
  Infection/fever, allergic symptoms, wheezing, upper/lower respiratory disease, gastrointestinal symptoms
Inflammation | 1 year
  Serum hs-CRP, Fibrinogen

CONTACTS AND LOCATIONS:
Overall Officials: Nikmah S Idris, MD, Principal Investigator — Indonesia University; Cuno SPM Uiterwaal, Ass Prof, MD, PhD, Study Chair — Julius Center; Sudigdo Sastroasmoro, Prof, MD, PhD, Study Director — CEEBM, University of Indonesia; Rulina Suradi, MD, Prof., Study Director — Indonesia University; Diederick E Grobbee, Prof, MD, PhD, Study Director — Julius Center; Mohammad Baharuddin, MD, Study Director — Budi Kemuliaan Hospital; Debby Bogaert, MD, PhD, Study Director — Utrecht University; Annemieke MV Evelein, MD, Principal Investigator — Julius Center; Wahyuni Indawati, MD, Principal Investigator — Indonesia University
Locations (1):
- Budi Kemuliaan Hospital, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Derived] Savitri AI, Idris NS, Indawati W, Saldi SR, Amelia D, Baharuddin M, Sastroasmoro S, Grobbee DE, Uiterwaal CS. BReastfeeding Attitude and Volume Optimization (BRAVO) trial: study protocol for a randomized controlled trial. Trials. 2016 Jun 2;17(1):271. doi: 10.1186/s13063-016-1397-y. PMID 27250730